CLINICAL TRIAL: NCT06111742
Title: Audiovisual Interactive Games to Improve Pediatric Patient Cooperation With Induction of Anesthesia and Alleviate Perioperative Anxiety
Brief Title: Audiovisual Interactive Games to Alleviate Pediatric Perioperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000033851; 000 (Other: CTGTY)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In the first phase (baseline measurement) neither participant nor investigator will be aware of the subjects group assignment. After this phase, due to the nature of the intervention, the experimental group will be aware they are in the intervention group when they see the gaming system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interactive Gaming Group (Experimental): Subjects will utilize an interactive gaming platform via the Bedside Entertainment and Relaxation Theater (BERT) directly prior to and during induction of anesthesia.
  Interventions: Device: Bedside Entertainment and Relaxation Theater (BERT)
- Standard of Care (No Intervention): Subjects will be offered standard of care interventions to improve preoperative anxiety. The interactive gaming system under investigation will not be available to this group.

INTERVENTIONS:
Device: Bedside Entertainment and Relaxation Theater (BERT) — BERT is a Nebula Capsule Max portable projector that creates a familiar theater experience designed for children to divert attention away from procedures. It is fitted with a remote control that can be utilized to manage on-screen activities. BERT can be used with any wall, ceiling, or projector screen to create the theater experience with a large screen. It can also be used with assist devices, such as steering wheel and noise-canceling headphones.
  Other Names: BERT
  Arms: Interactive Gaming Group

SUMMARY:
Pediatric anxiety upon induction of anesthesia is widely prevalent and can lead to negative patient psychological impact and hindrance to induction of anesthesia. Historically, premedication has been used as one means to improve pediatric preoperative anxiety and cooperation with induction. However, giving medication to children prior to surgery has drawbacks. Thus, other means have been proposed that may have similar benefits but fewer or different drawbacks. Recently, audiovisual distraction in the form of interactive games has been proposed. Such games have been in use at children's hospitals around the United States for more than five years. This study is a randomized trial that will explore using interactive games to improve pediatric perioperative anxiety in elective surgery compared with standard-of-care not including games. Perioperative anxiety with be evaluated using an observational scale.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 14 years of age;
* Undergoing non-emergent surgery at Yale New Haven Children's Hospital requiring general anesthesia;
* Chooses inhalational induction as induction method;
* Surgery qualified under one or more of the following fields: otolaryngology, ophthalmology, orthopedics, dentistry, gastrointestinal, general surgery

Exclusion Criteria:

* Altered mental status;
* Significant audiovisual deficits (per parent report and at discretion of study team);
* Received pharmacologic premedication

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Longhini, MD, Principal Investigator — Yale University School of Medicine, Department of Anesthesiology
Locations (1):
- Yale New Haven Children's Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data, in addition to study protocols, will be made available; the data will be made available on publication to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant randomized to experimental arm did not receive intervention
Groups:
- Healthcare Professionals: Health care providers' will be asked their opinions on the usefulness of AVG in reducing anxiety and the feasibility of such a program in a health care setting.
Period: Overall Study
Arm/Group | Interactive Gaming Group | Standard of Care | Healthcare Professionals
Started | 74 | 74 | 30
Child Participants | 37 | 37 | 0
Caretakers | 37 | 37 | 0
Completed | 71 | 74 | 30
Not Completed | 3 | 0 | 0
Not completed — Did not receive intervention | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interactive Gaming Group | Standard of Care | Healthcare Professionals | Total
Number analyzed (Participants) | 74 | 74 | 30 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Not collected for healthcare professionals.
  years
    Child participants: number analyzed (Participants) | 37 | 37 | 0 | 74
    Child participants | 7.35 (2.04) | 6.43 (1.98) |  | 6.89 (2.05)
    Caregivers: number analyzed (Participants) | 37 | 37 | 0 | 74
    Caregivers | 37.8 (6.1) | 37 (7) |  | 37.4 (6.07)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not collected for healthcare professionals.
  Participants
    Child Participants: number analyzed (Participants) | 37 | 37 | 0 | 74
    Child Participants: Female | 18 | 17 |  | 35
    Child Participants: Male | 19 | 20 |  | 39
    Caregivers: number analyzed (Participants) | 37 | 37 | 0 | 74
    Caregivers: Female | 29 | 32 |  | 61
    Caregivers: Male | 8 | 5 |  | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not collected for Caregivers or Healthcare Providers
  Participants
    number analyzed (Participants) | 37 | 37 | 0 | 74
    Hispanic or Latino | 13 | 13 |  | 26
    Not Hispanic or Latino | 21 | 24 |  | 45
    Unknown or Not Reported | 3 | 0 |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not collected for healthcare professionals or caregivers.
  Participants
    number analyzed (Participants) | 37 | 37 | 0 | 74
    American Indian or Alaska Native | 0 | 0 |  | 0
    Asian | 1 | 4 |  | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Black or African American | 7 | 5 |  | 12
    White | 26 | 25 |  | 51
    More than one race | 2 | 2 |  | 4
    Unknown or Not Reported | 1 | 1 |  | 2
Region of Enrollment [Number; unit: participants] — Population: Not collected for healthcare professionals or caregivers.
  participants
    United States: number analyzed (Participants) | 37 | 37 | 0 | 74
    United States | 37 | 37 |  | 74
Healthcare Professional Title [Count of Participants; unit: Participants] — Population: Only collected for healthcare professionals
  Participants
    Anesthesiologist: number analyzed (Participants) | 0 | 0 | 30 | 30
    Anesthesiologist | 0 | 0 | 5 | 5
    Anesthesiology Resident/Fellow: number analyzed (Participants) | 0 | 0 | 30 | 30
    Anesthesiology Resident/Fellow | 0 | 0 | 8 | 8
    Circulating Nurse: number analyzed (Participants) | 0 | 0 | 30 | 30
    Circulating Nurse | 0 | 0 | 6 | 6
    Certified Registered Nurse Anesthetist (CRNA): number analyzed (Participants) | 0 | 0 | 30 | 30
    Certified Registered Nurse Anesthetist (CRNA) | 0 | 0 | 3 | 3
    Scrub Technologist: number analyzed (Participants) | 0 | 0 | 30 | 30
    Scrub Technologist | 0 | 0 | 3 | 3
    Surgery Resident/Fellow: number analyzed (Participants) | 0 | 0 | 30 | 30
    Surgery Resident/Fellow | 0 | 0 | 5 | 5
Caregiver Relationship to Participant [Count of Participants; unit: Participants] — Population: Only collected for caregivers.
  Participants
    number analyzed (Participants) | 37 | 37 | 0 | 74
    Parent | 34 | 37 |  | 71
    Other | 3 | 0 |  | 3
Caregiver Surgical History, Previous Surgery [Count of Participants; unit: Participants] — Population: Only collected for caregivers.
  Participants
    number analyzed (Participants) | 37 | 37 | 0 | 74
    Yes | 23 | 28 |  | 51
    No | 14 | 9 |  | 23
Short State Anxiety Inventory Score at baseline [Mean (Standard Deviation); unit: score on a scale] — Score ranges from 6 to 24, higher scores suggest higher levels of anxiety. Population: Only collected for caregivers.
  score on a scale
    number analyzed (Participants) | 37 | 37 | 0 | 74
    (all) | 10.5 (5.3) | 11.4 (3.1) |  | 10.95 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Patient Anxiety Assessed by Modified Yale Perioperative Anxiety Score (mYPAS)
Description: The mYPAS is the gold standard for measuring pediatric perioperative anxiety. It is an observational-based 22-item instrument divided into five categories: activity, emotional expressivity, state of arousal, vocalization, and use of parents. The score ranges from 23 to 100, higher scores suggest higher levels of anxiety. It was developed at Yale University. This will be used for child participants only. Results presented here are mean change from baseline in anxiety during induction and upon Operating Room (OR) entry.
Time Frame: Baseline at OR entry (approximately 1 hour after baseline) and At Induction of Anesthesia (approximately 65 minutes after baseline),
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interactive Gaming Group | Standard of Care
Number analyzed (Participants) | 37 | 37
score on a scale
  Induction | 5 (18.3) | 21.4 (22.1)
  OR entry | 0.18 (9.7) | 8.9 (10.7)
Statistical Analysis 1: Comparison: Interactive Gaming Group vs Standard of Care; Induction; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Interactive Gaming Group vs Standard of Care; OR entry; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Mean Change in Caretaker Anxiety Assessed by Short State Anxiety Inventory Score
Description: The Short State Anxiety Inventory is a 6-item validated measure of anxiety in subjects aged 5 years and older. Subjects are asked to rate how they felt on a 4-point Likert scale in relation to feeling calm, tense, upset, relaxed, content, or worried. A score of 1 correlates to "not at all" and a score of 4 correlates to "very much." The final score is the sum of recorded values and ranges from 6 to 24, higher scores suggest higher levels of anxiety. This will be collected for caretakers only.
Time Frame: Baseline, After Induction of Anesthesia (approximately 1 hour after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interactive Gaming Group | Standard of Care
Number analyzed (Participants) | 37 | 37
score on a scale | -0.18 (3.20) | 1.89 (2.84)
Statistical Analysis 1: Comparison: Interactive Gaming Group vs Standard of Care; Test type: Superiority; p = 0.022, t-test, 2 sided

3. Secondary Outcome: Healthcare Professional Opinions on BERT Assessed With Health Professional Survey
Description: This survey will obtain health care providers' opinions on the usefulness of using the BERT system in reducing anxiety and the feasibility of such a program in a health care setting. Eligible individuals include: physicians, physician assistants/advanced practice providers, nurses, and other operating room staff.
Time Frame: During first 10 study days
Measure: Number; unit: percentage of participants
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 30
percentage of participants
  Rated BERT system "very favorable" or "favorable" for continued use | 97
  Believe system benefited children | 97
  Believe system benefited caregivers | 90
  Believe system benefited staff | 70
  Did not find system disruptive | 70

4. Secondary Outcome: Patient Induction Compliance Assessed by Induction Compliance Checklist
Description: The Induction Compliance Checklist is a validated 10-item observer-rated checklist of behaviors that interfere with induction of anesthesia. The score is the sum of the items checked. A perfect induction (the child does not exhibit negative behaviors, fear, or anxiety) is scored as 0, whereas the worst induction is a score of 9. A score greater than six is considered "poor" compliance. This will be collected for child participants only.
Time Frame: At Induction of Anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interactive Gaming Group | Standard of Care
Number analyzed (Participants) | 37 | 37
score on a scale | 1.0 (2.2) | 2.1 (2.5)
Statistical Analysis 1: Comparison: Interactive Gaming Group vs Standard of Care; Test type: Superiority; p = 0.046, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: up to one month
Arm/Group | Interactive Gaming Group | Standard of Care | Healthcare Professionals
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74 | 0/30
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT06111742/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT06111742/ICF_001.pdf